CLINICAL TRIAL: NCT05293626
Title: A Phase 1/2, Single-Arm, Open-Label, Dose-Finding Clinical Trial to Evaluate the Safety and Efficacy of Gene Therapy for Leber's Hereditary Optic Neuropathy (LHON) Associated With ND4 Mutation
Brief Title: Gene Therapy Clinical Trial for the Treatment of Leber's Hereditary Optic Neuropathy Associated With ND4 Mutations
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Neurophth Therapeutics Inc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NFS-01-US101
Record Dates: First submitted 2021-12-09; First posted 2022-03-24 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Leber Hereditary Optic Neuropathy (LHON)
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber | interventions — Needles; Syringes

STUDY DESIGN:
Intervention Model Description: 0.5E9 vg, 0.05 mL/eye/dose (low dose) 1.5E9 vg, 0.05 mL/eye/dose (starting dose) 3.0E9 vg, 0.05 mL/eye/dose (intermediate dose) 4.5E9 vg, 0.05 mL/eye/dose (high dose)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- NR082 injection (Experimental): Potential doses at the dose-finding stage:
  * 0.5E9 vg, 0.05 mL/eye/dose (low dose)
  * 1.5E9 vg, 0.05 mL/eye/dose (starting dose)
  * 3.0E9 vg, 0.05 mL/eye/dose (intermediate dose)
  * 4.5E9 vg, 0.05 mL/eye/dose (high dose)
  Interventions: Drug: NR082 Injection; Device: Injection needle

INTERVENTIONS:
Drug: NR082 Injection — The starting dose is 1.5E9 vg, 0.05 mL eye/dose.
  Dose Escalation:
  If drug-related dose-limiting toxicity (DLT) events are observed in ≤ 2 of the 6 evaluable subjects using the starting dose within 6 weeks after the dosing of NR082, the dose can be escalated to 4.5E9 vg, 0.05 mL eye/dose (high dose) after approval by SRC.
  Dose De-escalation： If drug-related dose-limiting toxicity (DLT) events are observed in > 2 of the 6 evaluable subjects using the starting dose within 6 weeks after the dosing of NR082, the dose can be de-escalated to 0.5E9 vg, 0.05 mL eye/dose (low dose) after approval by SRC.
  If drug-related dose-limiting toxicity (DLT) events are observed in > 2 of the 6 evaluable subjects within 6 weeks after the dosing of NR082 at the high dose, the dose can be de-escalated to 3.0E9 vg, 0.05 mL eye/dose (intermediate dose) after the approval by SRC.
Device: Injection needle — 19G 1 1/2IN TW filter needle with filter element (BD 305200)，used to NR082 Intraocular injection solution dose preparation; 30G 1/2IN injection needle (BD 305106)，used to NR082 Intraocular injection solution administration;
  1 ml screw top syringe (BD 309628),used to NR082 Intraocular injection solution dose preparation and administration.
  Other Names: Syringe

SUMMARY:
The objective of this clinical study is to evaluate the safety and efficacy of NR082 in the treatment of LHON caused by mitochondrial ND4 gene mutation. This study will enroll subjects aged ≥ 18 years old and ≤ 75 years old to receive a single unilateral intravitreal (IVT) injection of NR082 to evaluate its safety and efficacy. The clinical manifestations of all subjects are to be reduced visual acuity caused by LHON associated with ND4 mutation, with laboratory test showing G11778A mutation (a CLIA-certified laboratory) and reduced visual acuity lasted for > 6 months and < 10 years.

DETAILED DESCRIPTION:
At the dose-finding stage, the principle is that the Safety Review Committee (SRC) will decide whether to make dose adjustment based on the safety data of the starting dose. The starting dose is 1.5×109 vg, 0.05 mL eye/dose.The safety of the starting dose will be reviewed by the SRC, and dose escalation or de-escalation is by recommendation of the SRC.The safety of the starting dose will first be performed in 6 evaluable subjects.

Criteria for Dose Modification:

Dose Escalation:

If drug-related dose-limiting toxicity (DLT) events are observed in ≤ 2 of the 6 evaluable subjects within 6 weeks after the dosing of NR082 at the starting dose, the dose can be escalated to 4.5×109 vg, 0.05 mL eye/dose (high dose) after the approval by SRC.

Dose De-escalation:

If drug-related dose-limiting toxicity (DLT) events are observed in > 2 of the 6 evaluable subjects within 6 weeks after the dosing of NR082 at the starting dose, the dose can be de-escalated to 0.5×109 vg, 0.05 mL eye/dose (low dose) after the approval by SRC.

If drug-related dose-limiting toxicity (DLT) events are observed in > 2 of the 6 evaluable subjects within 6 weeks after the dosing of NR082 at the high dose, the dose can be de-escalated to 3.0×109vg, 0.05 mL eye/dose (intermediate dose) after the approval by SRC.

Enrollment Sequence:

* The enrollment sequence of any dose group (6 subjects) is that the 2nd subject and the 3rd subject will be enrolled at least 7 days after the enrollment of the 1st subject;
* The 4th, 5th and 6th subjects will be enrolled at least 7 days after the enrollment of the 2nd and the 3rd subjects.

The 7-day interval is to avoid acute safety events to the greatest possible extent

ELIGIBILITY:
Inclusion Criteria:

1. Age at the time of signing the informed consent form: the age of the subjects must be ≥ 18 years old and ≤ 75 years old.
2. The clinical manifested vision loss due to LHON, and any eye BCVA ≥ 0.5 LogMAR
3. The genotype testing result shows the presence of G11778A mutation in the ND4 gene, and the absence of the other primary LHON associated mutations in the mitochondrial DNA (mtDNA) (ND1 [G3460A] or ND6 [T14484C]) (confirmed by a CLIA-certified international laboratory
4. The vision loss in the eye with worse visual acuity lasted > 6 months and < 10 years at screening
5. Pupils can be adequately dilated for a thorough ocular examination and visual acuity test
6. Each eye of the subject must maintain at least Hand Motion VA (≤ 2.3 LogMAR) as defined in the ocular/vision examination manual (operating manual for refraction and VA examinations) in this study
7. Willingness to comply with the clinical study protocol and 5 years of long-term follow-up after administration
8. Male or female

   1. A male subject must agree to take contraceptive measures at least 6 months after the treatment visit;
   2. A female subject is eligible to participate if she is not pregnant , not breastfeeding, and at least one of the following conditions applies:i)Not a woman of childbearing potential (WOCBP) ;ii) A WOCBP who agrees to follow the contraception guidance for at least 6 months after the treatment visit
9. Written informed consent form must be obtained from the subject or his/her parent/legal guardian before any study-related procedures are performed.If the subject is legally blind (> 1.0 LogMAR or the readings of decimal visual acuity chart <0.1), an impartial witness must be present throughout the informed consent process and discussion process.

Exclusion Criteria:

1. Any known allergy and/or hypersensitivity to the study drug or its constituents
2. Contraindication to IVT injection in any eye
3. IVT drug delivery to any eye within 30 days prior to the screening visit
4. History of vitrectomy in either eye
5. Narrow anterior chamber angle in any eye contra-indicating pupillary dilation
6. Presence of disorders or diseases of the eye or adnexa, excluding LHON, which may interfere with visual or ocular assessments, including spectral-domain optical coherence tomography (SD-OCT), during the study
7. Presence of known/documented mutations, other than the LHON-related mutation, which are known to cause pathology of the optic nerve, retina or afferent visual system
8. Presence of systemic or ocular/vision diseases, disorders, or pathologies, other than LHON, known to cause or be associated with vision loss, or whose associated treatment(s) or therapy(ies) is/are known to cause or be associated with vision loss
9. Presence of optic neuropathy from any cause other than LHON
10. Presence of illness or disease that, in the opinion of the investigator, include symptoms and/or the associated treatments that can alter visual function, for instance cancers or pathology of the central nervous system (CNS), including multiple sclerosis (diagnosis of multiple sclerosis must be based on the 2010 Revisions to the McDonald Criteria) , and/or diseases or conditions that affect the safety of subjects participating in the study
11. History of recurrent uveitis (idiopathic or immune-related) or active ocular inflammation
12. Participated in another clinical study and receive an IMP within 90 days prior to the screening visit

    a) Exceptions: Subjects who have completed the clinical study of idebenone as IMP > 90 days prior to the screening visit and has completely discontinued idebenone at least 7 days prior to dosing are still eligible to participate in the study.
13. Any eye has previously received ocular gene therapy
14. Subjects who refused to stop using idebenone
15. Have undergone ocular surgery of clinical relevance (per investigator's assessment) within 90 days prior to the screening visit
16. Female subjects who are breastfeeding or plan to breastfeed within the first 6 months after the administration of NR082 Injection
17. History of drug or alcohol abuse (including heavy smoking, i.e., > 20 cigarettes per day or >20 pack-years [equivalent to one pack a day for 20 years or 2 packs a day for 10 years])
18. Human immunodeficiency virus (HIV) antibody, syphilis antibody and HCV antibody positive are excluded; hepatitis B test that shows a clinically significant active infection requiring treatment (defined as the presence of hepatitis B core antibody [HBcAb] positive or hepatitis B surface antigen [HBsAg] positive, and hepatitis B virus deoxyribonucleic acid [HBV-DNA]) > 1000 copies/mL or according to local laboratory method above lower limit of quantitative detection) are excluded
19. Unable to tolerate (e.g., immunomodulatory regimen) or unable or unwilling to comply with all the protocol requirements
20. Subjects from the study site fail to comply with or do not agree to comply with local and institutional guidelines for suspected 2019 novel coronavirus (COVID-19) infection/testing
21. Any other exclusions determined by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | 52 weeks
  Incidence of adverse events (AEs) within 52 weeks of NR082 intravitreal injection at different doses
Incidence of serious adverse events (SAEs) | 52 weeks
  Incidence of serious adverse events (SAEs)within 52 weeks of NR082 intravitreal injection at different doses
Incidence of dose-limiting toxicities (DLT) | 52 weeks
  Incidence of dose-limiting toxicities (DLT) (ocular and non-ocular) within 52 weeks of NR082 intravitreal injection at different doses

SECONDARY OUTCOMES:
Proportion (percent) of subjects with an improvement of ≥ 0.3 LogMAR from baseline in Best corrected visual acuity(BCVA) in the study eye | At Weeks 2, 6,12, 26, 40, 52, 78, 104, 156, 208, and 260
  ETDRS visual acuity charts will used to assess proportion (percent) of subjects with an improvement of ≥ 0.3 LogMAR from baseline in Best corrected visual acuity(BCVA)
Mean change from baseline in BCVA (LogMAR) in the study eye | At Weeks 2, 6,12, 26, 40, 52, 78, 104, 156, 208, and 260
  ETDRS visual acuity charts will used to assess mean change from baseline in BCVA (LogMAR)
Mean change in BCVA (LogMAR) compared to nadir* | At Weeks 2, 6,12, 26, 40, 52, 78, 104, 156, 208, and 260
  ETDRS visual acuity charts will used to assess mean change in BCVA (LogMAR) compared to nadir
Change from baseline in thepattern standard deviation (PSD)in the study eye | At Weeks 2, 6,12, 26, 40, 52, 78, 104, 156, 208, and 260
  Visual field parameters will evaluate alterations in function of different region the retina. The HVF analyzer is used to perform standard automated perimetry, and the kinetic visual field is measured by the Humphrey static visual field automatically detected by the computer, including the foveal and macular thresholds, as well as the central field. Change from baseline in thepattern standard deviation (PSD)in the study eye.
Change from baseline in the visual field index (VFI) in the study eye | At Weeks 2, 6,12, 26, 40, 52, 78, 104, 156, 208, and 260
  Visual field parameters will evaluate alterations in function of different region the retina. The HVF analyzer is used to perform standard automated perimetry, and the kinetic visual field is measured by the Humphrey static visual field automatically detected by the computer, including the foveal and macular thresholds, as well as the central field. Change from baseline in the visual field index (VFI) in the study eye.
Change from baseline in the mean deviation (MD) in the study eye | At Weeks 2, 6,12, 26, 40, 52, 78, 104, 156, 208, and 260
  Visual field parameters will evaluate alterations in function of different region the retina. The HVF analyzer is used to perform standard automated perimetry, and the kinetic visual field is measured by the Humphrey static visual field automatically detected by the computer, including the foveal and macular thresholds, as well as the central field. Change from baseline in the mean deviation (MD) in the study eye.
Change from baseline in spatial frequency parameters of contrast sensitivity in the study eye | At Weeks 2, 6,12, 26, 40, 52, 78, 104, 156, 208, and 260
  The contrast sensitivity examination measures the subject's ability to discern targets presented at varying spatial frequencies or sizes under different contrast levels. The contrast sensitivity examination measures the full range of visual sensitivity, including brightness and contrast, and it may be used as a comprehensive assessment of visual function
Change from baseline in visual evoked potential (VEP) parameters in the study eye | At Weeks 2, 6,12, 26, 40, 52, 78, 104, 156, 208, and 260
  VEP is a visual electrophysiological examination used to identify possible ischemic optic neuropathy,including the P100 Latency,P100 Amplitude,P2 Latency,P2 Amplitude.
To evaluate immunogenicity | At Weeks 1, 2, and 6
  A central laboratory will be used to evaluate anti-AAV2 neutralizing antibodies in the serum samples of all subjects.These samples will be tested by the sponsor or its designee to detect anti-AAV2 neutralizing antibodies in the samples and report the titer of confirmed positive samples. Samples confirmed positive for anti-AAV2 neutralizing antibodies will also be evaluated for the presence of neutralizing antibodies.
To evaluate immunogenicity | At Weeks 1, 2, 6, 12, 26, 40, and 52
  The interferon gamma enzyme-linked immunospot (ELISpot) assay will be performed to measure the proliferative response of lymphocytes to AAV2 antigen and ND4 peptide.The number of activated cells in the sample was calculated.
To evaluate vector shedding | At Weeks 1, 2, 6, 12, 26, 40, and 52
  Assessment of vector DNA shedding in tears (both eyes).Samples were analyzed to determine the presence of viral DNA in tears .
To evaluate biodistribution | At Weeks 1, 2, 6, 12, 26, 40, and 52
  Assessment of biodistribution in whole blood.Samples were analyzed to determine the presence of viral DNA in whole blood.
To evaluate the improvement in BCVA of the study eye (< 0.3 LogMAR) | At Weeks 52, 78, 104, 156, 208, and 260
  ETDRS visual acuity charts will used to assess proportion (percent) of subjects with an improvement of ≥ 0.2 LogMAR and ≥ 0.1 LogMAR from baseline in BCVA Proportion (percent) of subjects with visual acuity of > 1.0 LogMAR before and after treatment
To evaluate the change from baseline in VFQ-25 | At Weeks 2, 26, 52, 104, 156, 208, and 260
  VFQ-25 is a 25-item short form version of the 51-item National Eye Institute Visual Function Questionnaire (NEI VFQ), which can effectively measure patient-reported outcomes (including quality of life, QoL).It consists of 25 items from 12 dimensions. The total score and the score of each dimension are the mean values of non-missing items of corresponding dimensions or items, with the score range from 0 to 100 , higher scores mean a worse outcome.
To evaluate the change from baseline in quality of SF-36 | At Weeks 2, 26, 52, 104, 156, 208, and 260
  The SF-36 questionnaire is a universal tool for evaluating patient-reported QoL outcome. SF-36 comprises 36 questions which cover eight domains of health: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions. The scale score of each domain will be calculated based on the total score of the items included in the said domain and re-adjusted to 0-100,higher scores mean a worse outcome.
Change from baseline in retinal nerve fiber layer (RNFL) thickness of the study eye | At Weeks 2, 6,12, 26, 52, 104, 156, 208, and 260
  OCT is an imaging technology to investigate the ocular fundus by using of the basic principle of low-coherence light interferometry. It detects the reflection or diffusion signals of biological tissue layers of different depths by inputting low-coherence light and obtains the images and quantitative results of the microscopic structure of the retina
Change from baseline in retinal ganglion cell complex thickness of the study eye | At Weeks 2, 6,12, 26, 52, 104, 156, 208, and 260
  OCT is an imaging technology to investigate the ocular fundus by using of the basic principle of low-coherence light interferometry. It detects the reflection or diffusion signals of biological tissue layers of different depths by inputting low-coherence light and obtains the images and quantitative results of the microscopic structure of the retina
To evaluate the visual function improvement after NR082 treatment | At Weeks 2, 6,12, 26, 52, 104, 156, 208, and 260
  Early Treatment Diabetic Retinopathy Study(ETDRS) visual acuity charts will used to assess proportion (percent) of subjects with an improvement of ≥ 0.3 LogMAR from baseline in Best corrected visual acuity(BCVA) of the non-study eye

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Stanford Byers Eye Institute, Palo Alto, California
  - University of Colorado Health Eye Center, Aurora, Colorado
  - Wills Eye Hospital, Neuro Ophthalmology Department, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No